CLINICAL TRIAL: NCT06286904
Title: Sleep Position Pattern Recording - A Validation Study
Brief Title: Sleep Position Pattern Recording
Status: Not yet recruiting | Type: Observational
Sponsor: Myant Medical Corp. (Industry)
Collaborators: McMaster University (Other)
Responsible Party: Sponsor
Other Study IDs: McMaster-Myant 16633
Record Dates: First submitted 2024-02-16; First posted 2024-02-29 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Pregnant Women
Keywords: sleep; wearable electronic devices; Pregnant Women; Posture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sleep position detection: Accuracy of Skiin Garment system for detecting sleep position of pregnant womem.
  Interventions: Device: Skiin Garment system

INTERVENTIONS:
Device: Skiin Garment system — Individuals will be asked to wear a Skiin Garment system for the duration of their hospitalization (minimum one day).The system will collect accelerometer, ECG, temperature, heart rate, steps and sleep metrics data if enable. Then, they will be asked to answer a questionnaire about their experiences with the device and the study.

SUMMARY:
The main goal of this study is to validate the accuracy of the body position detection by non-invasive wearable monitors (Skiin garments, Myant Medical Corp) during sleep in pregnant participants. This is a first step towards examining the association between maternal sleep position and fetal growth.

DETAILED DESCRIPTION:
Individuals who are eligible to the study and provided consent to participate will be asked to:

1. Wear the Skiin Garment system for the duration of their time in the hospital (minimum 1 nights until they are discharged from hospital).
2. Complete a study completion questionnaire about their experience with the device and the study.

The Skiin Garment system is composed by biosensing garments presented in different form factors (bra, chest band, or underwear). It captures physiological metrics and relay information from a pod to local hub with Bluetooth.

The true body position will be obtained using visual observations and cameras.

ELIGIBILITY:
Inclusion Criteria:

* Assigned female at birth
* Currently pregnant
* Admission to MUMC Antenatal Clinic with anticipation of being admitted for greater than 24 hours
* Able and willing to provide informed consent to participate

Exclusion Criteria:

* Unestablished gestational dating (based on first-trimester ultrasound)
* Known maternal cardiac or pulmonary disorder
* Known sleep disorders (i.e., sleep apnea, periodic limb movement disorder, etc.)
* Known fetal chromosomal or structural abnormalities
* Known highly sensitive skin/skin sensitivities to textile electrodes

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — This study will enroll pregnant women.
Study Population: Pregnant women admitted in the antenatal in-patient clinic at McMaster University Medical Centre for greater than 24 hours.
Sampling Method: Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Skiin Garment system for detecting sleep position of pregnant women | Recorded during the night, during 6 to 8 hours.
  Sleep position will be identified through the Skiin Garment system via accelerometry, and compared to visual confirmation of sleep position.

SECONDARY OUTCOMES:
Questionnaire on wearable device invasiveness and satisfaction | One time point, on the morning after one night wearing the Skiin Garment system
  Pregnant women will be asked to answer a questionnaire at the end of their participation in the study. It contains questions related to patients' experience wearing the Skiin Garment system, including invasiveness and satisfaction.
  This is an ad-hoc questionnaire titled "SPV_Satisfaction_Questionnaire_v1_2023-04-03" containing 20 questions: 14 questions use a Likert scale design, 3 questions are single choice answer, and 3 questions are open-ended questions. Results are not reported as a total score on a scale but descriptive statistics will be used individually per question.
Participant recruitment rate | From the beginning to the end of the recruitment, up to 1 year.
  Recruitment rate will be calculated as the number of participants who consent to participant divided by the number of participants who consent to be contacted.
Participant retention rate | From the beginning to the end of participation, up to 1 year.
  The retention rate will be calculated as the number of participants who remain in the study divided by the number of participants who initially consent to participate.

CONTACTS AND LOCATIONS:
Overall Officials: Eran Ashwal, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No